CLINICAL TRIAL: NCT05861479
Title: Assessment of the Prognostic Value of the Estimation of Plasma Volume or Its Variation in Patients With Pulmonary Arterial Hypertension (PAH) or Chronic Thromboembolic Pulmonary Hypertension (CTEPH) After Acute Right Heart Failure
Brief Title: Prognostic Value of Estimated Plasma Volume in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI167
Record Dates: First submitted 2023-05-05; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Acute Right Heart Failure
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the prognostic value of the estimation of plasma volume or its variation in patients with pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH) after acute right heart failure.

DETAILED DESCRIPTION:
The aim of the study is to show that a low plasma volume status, assessed by the Strauss (estimated plasma volume variation) and the Duarte (instantaneous estimated plasma volume) formulas evaluated during acute right heart failure in patients presenting with PAH or CTEPH, is associated with better long-term outcomes.

Optimization of plasma volume is important for patients with PAH and CTEPH and constitutes a prognostic factor. However, plasma volume status can be difficult to assess in clinical practice. Different formulas have been developed and have shown interest in patients with congestive heart failure with an association between plasma volume estimation and long-term prognosis.

Acute right heart failure may occur in patients with PAH and CTEPH. Thus, the investigators plan to study the prognostic value of these formulas evaluating plasma volume, in patients with PAH or CTEPH, after acute right heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of PAH or CTEPH, referred to the medical department of the investigators
2. Patient with acute right heart failure defined by at least 2 of the following clinical features: worsening of peripheral oedema, development or increase of ascites, weight gain of more than 2.5 kg in 1 week preceding the visit and decline in one NYHA functional class compared to the previous stable state

Exclusion Criteria:

1) Patients with another cause of pulmonary hypertension than PAH or CTEPH, either groups 2, 3 or 5 of the current clinical classification of pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients with idiopathic, heritable, drug-induced, connective tissue disease-associated, porto-pulmonary or HIV-associated disease were enrolled. At the diagnosis visit, mean±SD age was 59±12 years, 56% of the patients were women and most patients were in World Health Organization/New York Heart Association (WHO/NYHA) Functional Class III or IV.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Survival | From the first visit to 1st April 2023
  Death
Recurrence of acute right heart failure | From the first visit to 1st April 2023
  Hospital admission for acute right heart failure
Acute right heart failure-free survival | From the first visit to 1st April 2023
  First event: death or hospital admission for acute right heart failure

IPD SHARING:
Plan to Share IPD: Undecided